CLINICAL TRIAL: NCT05673395
Title: Effects of Alkaline-reduced Water Generated From Electrolyzed Device (CGM MWPI-2101) on High-intensity Exercise-induced Oxidative Stress and Fatigue in Young Male Healthy Adults: Controlled, Randomized, Double-blind Clinical Trial
Brief Title: Drinking Effect of Electrolyzed Alkaline Reduced Water on Oxidative Stress and Fatigue After Intense Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyu Jae Lee (Other)
Collaborators: Ceragem Inc. (Industry)
Responsible Party: Sponsor-Investigator, Kyu Jae Lee, Professor, Wonju Severance Christian Hospital
Organization: Wonju Severance Christian Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: EMB-2022-02
Record Dates: First submitted 2022-12-19; First posted 2023-01-06 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Oxidative Stress

STUDY DESIGN:
Intervention Model Description: The participants were randomly divided into two groups (n = 12) according to the sequence of random numbers obtained through an online number generator. After the first clinical trial, A wash-out period of one week was applied to prevent carry-over before crossing over, and the second clinical trial was performed.
Who Masked: Participant, Investigator
Masking Description: double blind (participants, investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EARW group (Experimental): This group drink electrolyzed alkaline reduced water (EARW, pH 9.5) 10 mL/kg body weight in 10 min after exercise.
  Interventions: Device: Electrolyzed alkaline reduced water generator
- PW group (Sham Comparator): PW is purified water generated from sham device, and PW group drink 10 mL/kg body weight in 10 min after exercise.
  Interventions: Device: Electrolyzed alkaline reduced water generator

INTERVENTIONS:
Device: Electrolyzed alkaline reduced water generator — Participants drink water (10 mL/kg body weight) generated from the device after intensive excercise.
  Other Names: Electrolyzed alkaline ionizer (CGM MWPI-2101

SUMMARY:
The goal of this clinical trial is to test the drinking effect of electolyzed alkaline reduced water (ARW) generated from alkaline ionizer (CGM MWPI-2101) on oxidative stress and fatigue after high-intensity exercise in healthy people. The main question[s] it aims to answer are:

* [question 1] Can pH 9.5 EARW reduce oxidative stress compared to purified water (PW)
* [question 2] Can pH 9.5 EARW decrease fatigue markers in blood

Participants will drink water from the experimental device after high-intensity exercise. Blood sample will be collected before exercise, after highly intensive exercise, and after then 15 min. of drinking water.

Researchers will compare EARW group and PW group to see the anti-oxidative and anti-fatigue effects.

DETAILED DESCRIPTION:
This study was designed as a randomized, controlled, crossover, double-blind clinical trial with a single intervention of ARW intake (pH 9.5, 10 mL/kg body weight) after highly intense exercise.

The participants were divided into two groups, wherein they consumed either puriﬁed water (PW group) or EARW (EARW group). Blood samples were collected before exercise, immediately after exercise, and 15 min after drinking water.

For the anti-oxidative effect, ROS, NO, GPx, and MDA levels were measured. For the anti-fatigue effect, latate, lactate dehydrogenase, phosphate and calcium were measured.

ELIGIBILITY:
Inclusion Criteria:

* healthy male participants aged 19-25 years
* physically active with a normal body mass index (BMI)
* had not smoked for 3 months or consumed alcohol for more than a week prior to the start of the study.

Exclusion Criteria:

* any kind of visible or known disease
* hypertension,
* musculoskeletal injuries in the previous three months,
* breathing difﬁculties,
* metabolic diseases,
* autoimmune disease,
* rash,
* urticaria.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
EARW consumption is effective in reducing oxidative stress | 15 minutes
  Reactive oxygen species, nitric oxide, glutathione peroxidase, malondialdehyde

SECONDARY OUTCOMES:
The effects of EARW consumption on exercise-induced fatigue markers in healthy young adults | 15 minutes
  Lactate levels, phosphate levels, cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Jae Lee, Ph.D., Study Chair — 20, Ilsan-dong, Wonju, Gangwon-do, South Korea, 26426
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Ganwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No